CLINICAL TRIAL: NCT05176431
Title: Comparation of Radial and Focused Extracorporeal Shock Wave Therapies According to Age and Body Mass Index in the Treatment of Coccydynia.
Brief Title: Radial and Focused ESWT in the Treatment of Coccydynia According to Age and Body Mass Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Volkan Şah, Principal Investigator, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: University of Yuzuncu Yil
Record Dates: First submitted 2021-11-30; First posted 2022-01-04 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Coccyx Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Focused extracorporeal shock wave therapy (Active Comparator)
  Interventions: Device: ESWT (wave type: focused)
- Radial extracorporeal shock wave therapy (Active Comparator)
  Interventions: Device: ESWT (wave type: radial)
- Sham extracorporeal shock wave therapy (Sham Comparator)
  Interventions: Device: ESWT (wave type: sham)

INTERVENTIONS:
Device: ESWT (wave type: focused) — Extracorporeal Shock Wave Therapy, device: Electronica, Pagani, Italy
  Arms: Focused extracorporeal shock wave therapy
Device: ESWT (wave type: radial) — Extracorporeal shock wave therapy, device: Electronica, Pagani, Italy
  Arms: Radial extracorporeal shock wave therapy
Device: ESWT (wave type: sham) — Extracorporeal shock wave therapy, device: Electronica, Pagani, Italy
  Arms: Sham extracorporeal shock wave therapy

SUMMARY:
To date, focused and radial types of ESWT have been effectively used in the treatment of coccydynia. However, studies directly addressing a comparison between radial and focused types of ESWT in coccydynia have not been done. Therefore, this study aims to evaluate comparative effects of radial and focused ESWT options on coccydynia.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of coccydynia by clinical examination and X-ray imaging.
* be aged ≥18 at the time of diagnosis
* be give informed consent

Exclusion Criteria:

* Malignancy
* Those who have received ESWT treatment before
* Pediatric patients
* Patients with infection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 1 minute
  pain evaluation, higher scores mean a worse outcome.
Oswestry Disability Index | 5 minutes
  functional status of low back pain, higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Yuzuncu Yil University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No